CLINICAL TRIAL: NCT01812889
Title: A Two Part Randomized, Open-Label Phase I Safety and Pharmacokinetic Evaluation of Gel and Ovule Formulations of TOL-463 (Intravaginal Therapy) in 18-45 Year Old Healthy Female Subjects and Women With Vaginitis
Brief Title: Evaluation of Intravaginal Gel and Ovule Formulations of TOL-463
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-0077; HHSN272200800024C; TOL-463
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Vaginal Infection
Keywords: bacterial vaginosis, vulvovaginal candidiasis, TOL-463, intravaginal therapy, vaginitis, women, cross-over
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Candidiasis, Vulvovaginal

ARMS (2):
- Part 2 (Active Comparator): 10 women diagnosed with BV, 10 diagnosed with VVC will be randomized to receive either TOL-463 gel or TOL-463 ovules administered intravaginally once daily for 7 consecutive days
  Interventions: Drug: TOL-463 Vaginal ovule; Drug: TOL-463 Vaginal gel
- Part 1 (Active Comparator): 20 Healthy women randomized, two-way crossover design will receive a single dose of TOL-463 gel and ovule intravaginally, separated by a minimum of 7 day washout period between administrations
  Interventions: Drug: TOL-463 Vaginal ovule; Drug: TOL-463 Vaginal gel

INTERVENTIONS:
Drug: TOL-463 Vaginal ovule — TOL-463 Vaginal Ovule
Drug: TOL-463 Vaginal gel — TOL-463 Vaginal Gel

SUMMARY:
The purpose of this study is to determine the safety, local tolerability and pharmacokinetic parameters of TOL-463 intravaginal dosage forms in both healthy, nonpregnant females following single dose administration (Part 1), and in nonpregnant women with vaginitis following multi-dose administration (Part 2).

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety, local tolerability and pharmacokinetic parameters of TOL-463 intravaginal dosage forms in both healthy, nonpregnant females following single dose administration (Part 1), and in nonpregnant women with vaginitis following multi-dose administration (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Adult women of any race between 18 to 45 years of age (inclusive).
* Subjects must be able to give voluntary written informed consent before any study related procedure is performed.
* Subjects must have a negative serum pregnancy test at Screening and negative urine pregnancy test at all other clinical site visits, as applicable.
* Subjects either have no childbearing potential (as defined below) (Note 1) or agree to avoid becoming pregnant from the day of screening through one month after the last study Day using one of the following acceptable methods of birth control (Note 2) in addition to the use of non-lubricated condoms by the male partner (even if vasectomized).

  * Hormonal contraceptives
  * Abstinence
  * Note 1: Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy or status after hysterectomy.
  * Note 2: Intravaginal or intra-uterine contraceptives and contraceptive devices (IUDs) are not acceptable forms of birth control for this study.
* Subjects must agree to refrain from douching or using any intravaginal products (i.e., contraceptive creams, gels, foams, sponges, lubricants, etc.) or IUDs during the study period.
* Subjects must agree not to donate blood during the study and up to 14 days after the end of the study.
* Subjects willing and able to comply with all study requirements.

For Part 1 Only

* Subjects must be healthy as determined by medical history, physical examination, vital signs, pelvic examination and laboratory evaluations (hematology, clinical chemistry and urinalysis tests) within study-defined ranges at Screening.
* Subjects must be without current symptomatic or asymptomatic bacterial vaginosis, candida vulvovaginitis or any other form of vaginitis by clinical and microbiologic testing.
* Subjects must be willing to abstain from sexual intercourse for 24 hours prior to each site visit.

For Part 2 Only

* Subjects with vaginitis must be otherwise healthy based on medical history, physical examination, vital signs, pelvic examination and laboratory evaluations (hematology, clinical chemistry and urinalysis tests) within study-defined ranges at Screening.
* Subjects with vaginitis must be willing to abstain from sexual intercourse 24 hours prior to the first dose of study medication and throughout the last visit of the study.

Exclusion Criteria:

* A history of clinically significant acute illness (resolved within 4 weeks of screening) or any other condition which, in the opinion of the Site Principal Investigator (PI), would jeopardize the safety of the subject or impact the validity of the study results.
* Subjects with intrauterine devices.
* Subjects with renal dysfunction (serum creatinine >/= 1.2 mg/dL).
* Subjects with underlying metabolic or endocrine dysfunction, such as diabetes mellitus, Cushing's disease, Addison's disease, or hypo- or hyperthyroidism.
* Subjects who test positive for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
* Subjects who have diseases known to cause immunodeficiency, e.g., AIDS, advanced malignancy, anemia or severe vitamin deficiency.
* Subjects who test positive for Trichomonas vaginalis, Neisseria gonorrhea, or Chlamydia trachomatis at screening.
* Subjects with active genital lesions at screening, including syphilitic chancre, herpetic lesions, or genital warts (HPV).
* Subjects who have had major surgery within 4 weeks of screening.
* Subjects with an uncontrolled active illness (e.g., active infection) or fever (oral temperature >/=100 degrees F or >/= 37.7 degrees C) at screening.
* Subjects with a known sensitivity to any ingredient in TOL-463 vaginal gel or ovule.
* With the exception of oral contraceptives, use of a prescription medication, notably antimicrobial agents, corticosteroids or other immuno-suppressants, within 14 days prior to Day 1 of study treatment, unless in the opinion of the PI, the substance would not likely impact the conduct or results of this study.
* Subjects with any current unstable medical condition(s) requiring prescription medication(s) that would preclude accurate evaluation of subjects or otherwise impact the conduct or results of the study.
* Subjects who have received an investigational drug in a clinical trial within 30 days prior to screening.
* Women who are pregnant or breast feeding. Subject has a positive history for alcohol abuse or dependence and/or a positive urine screen test for alcohol and drugs of abuse [amphetamines, barbiturates, benzodiazepines, cocaine metabolites, marijuana, opiates, phencyclidine (PCP)] at screening or at any check-in prior to receiving study drug.
* Subjects who have donated blood within the past 30 days prior to Day 1 of treatment with study drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The local (vulvovaginal) and systemic safety and tolerability of TOL-463 gel and ovules following a single intravaginal administration in healthy female subjects and following daily dosing for 7 days in women with BV or VVC will be assessed. | Following daily dosing for 1 or 7 days
Adverse events (AEs) will be monitored throughout the course of the study following administration of Investigational Product (IP). | Up to Day 16

SECONDARY OUTCOMES:
Standard PK parameters (half-life, Cmax, Tmax and AUC), will be assessed following single-dose administration of TOL-463 gel and ovule in healthy subjects and after single- and multiple-dose administration of TOL-463 gel or ovules in women with BV or VVC | Once daily for 1 or 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States